CLINICAL TRIAL: NCT07050056
Title: Tislelizumab Combined With Thoracic Radiotherapy as Neoadjuvant Therapy for Resectable NSCLC: A Single Arm, Phase II Clinical Study
Brief Title: Tislelizumab Combined With Thoracic Radiotherapy as Neoadjuvant Therapy for Resectable NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Buhai Wang, Executive Vice-President, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ky220
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Resectable NSCLC
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab plus radiotherapy (Experimental): Tislelizumab IV 200mg, d1, Q3W; concurrently combined with 40Gy/20f radiotherapy (3D-CRT/IMRT, IMRT, targeting only the lesion and positive lymph nodes), for 3-4 cycles.
  Interventions: Drug: Tislelizumab; Radiation: 3D-CRT/IMRT

INTERVENTIONS:
Drug: Tislelizumab — 200mg, iv, Q3W, 3-4 cycle
Radiation: 3D-CRT/IMRT — 40Gy in 20 fractions

SUMMARY:
This study aims to explore the efficacy and safety of radiotherapy combined with immunotherapy in the neoadjuvant treatment of resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form (ICF);
* Aged 18-70 years, regardless of gender;
* Previously untreated, histologically confirmed resectable stage IB-IIIA NSCLC (AJCC 9th edition staging);
* At least one measurable lesion per RECIST v1.1 criteria;
* Willing to provide PD-L1 immunohistochemistry slides and corresponding pathology reports for biomarker evaluation;
* Presence of lesions suitable for radiotherapy as assessed by the study team;
* ECOG performance status of 0-1;
* Adequate organ function;
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures;
* Sufficient pulmonary function to tolerate planned lung resection surgery, as assessed by a surgeon;
* Women of childbearing potential must have a negative serum pregnancy test within 3 days prior to the first dose. Both female participants of childbearing potential and male participants with partners of childbearing potential must agree to use highly effective contraception during the study and for 180 days after the last dose of the study drug.

Exclusion Criteria:

* Presence of locally advanced unresectable or metastatic disease;
* NSCLC involving the superior sulcus, large cell neuroendocrine carcinoma (LCNEC), or sarcomatoid tumors;
* Participants with known EGFR mutations or ALK translocations (non-squamous NSCLC subjects must have confirmed EGFR/ALK mutation status);
* Prior systemic anticancer therapy for early-stage NSCLC, including investigational drugs; Contraindications to radiotherapy or inability to undergo radiotherapy;
* History of (non-infectious) pneumonitis/interstitial lung disease requiring steroids or current pneumonitis/interstitial lung disease requiring steroid treatment;
* Known active tuberculosis (TB) history; Known active infection requiring systemic therapy; Any known or suspected autoimmune disease or immunodeficiency;
* Active hepatitis B infection; Administration of live vaccines within 30 days before the first dose;
* Grade ≥2 peripheral neuropathy;
* Prior treatment with PD-1/PD-L1 inhibitors or drugs targeting other T-cell receptors (e.g., CTLA-4, OX-40, etc.);
* History of severe hypersensitivity to monoclonal antibodies;
* Severe or uncontrolled underlying medical conditions;
* Any condition that, in the investigator's judgment, may confound study results, interfere with the subject's participation, or compromise the subject's best interest in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 18 months
  Complete pathological response (pCR), defined as the proportion of patients in the ITT analysis set and surgical population analysis set who have no residual tumor in the resected primary tumor and metastatic lymph nodes as assessed by the investigator after the completion of neoadjuvant therapy. Patients who do not meet these criteria, including those who do not undergo surgical resection, will be considered non-responders.

SECONDARY OUTCOMES:
MPR Rate | 18 months
  Major pathological response (MPR) was defined as the proportion of patients in the ITT analysis set and surgical population analysis set with ≤ 10% residual viable tumor cells in the resected primary tumor and metastatic lymph nodes after the completion of neoadjuvant therapy as assessed by the investigator. Patients who do not undergo surgical resection for reasons such as disease progression will be considered non-responders.
1-year EFS Rate | Baseline up to 1 years
  1-year EFS rate is defined as the proportion of patients who have not experienced radiographic disease progression, local recurrence or distant metastasis, or death due to any cause assessed by the investigator according to RECIST 1.1 Version, from enrollment to 1 year in the intent-to-treat (ITT) analysis set. The 1-year EFS rate is evaluated by the Kaplan-Meier (KM) method.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Northern People Hospital, Yangzhou, Jiangsu, China